CLINICAL TRIAL: NCT06635278
Title: Effect of Mindfulness Meditation on Perceived Stress, Somatic Symptoms and Inflammatory Biomarkers Among Nurses
Brief Title: Mindfulness Meditation: Alleviating Symptoms and Inflammation in Nurses
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hossam Najjem Alhawatmeh, Associate Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/319
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Inflammation; Somatization
Keywords: Mindfulness Meditation; Nurses; Somatic symptoms; Leptin; Interleukin-6; Tumor necrosis factor- alpha; Perceived stress
MeSH Terms: conditions — Inflammation; Medically Unexplained Symptoms | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the participants' group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurses receiving mindfulness meditation (Experimental): The experimental group received eight 60-minute weekly sessions of mindfulness meditation over eight weeks in a private and quiet room at the hospital, according to Smith's (2005) recommendation. The theory-based program (Smith, 2005) includes the ABC standardized versions of MBI (Smith, 2005), described as follows:
  * Body sense meditation
  * Rocking meditation
  * Breathing meditation
  * Mentra meditation
  * Visual Image meditation
  * External image meditation
  * Meditation of a sound
  * Open monitoring (Mindfulness) meditation
  Interventions: Behavioral: Mindfulness meditation
- Nurses will receive no intervention or materials from the experimenter (No Intervention): Control group will receive a traditional care provided usually for patients in the hospital

INTERVENTIONS:
Behavioral: Mindfulness meditation — The experimental group received eight 60-minute weekly sessions of mindfulness meditation over eight weeks in a private and quiet room at the hospital, according to Smith's (2005) recommendation. The study intervention was an audio based MBI sent to them by the WhatsApp application. It is a free, self-paced program developed by a study researcher based on the Smith's (2005) protocol.
  The theory-based program (Smith, 2005) includes the ABC standardized versions of MBI (Smith, 2005), described as follows:
  * Meditation of the body (Body sense meditation)
  * Meditation of the body (Rocking meditation)
  * Meditation of the body (Breathing meditation)
  * Meditation of mind (Mentra meditation)
  * Meditation of mind (visual Image)
  * Meditation of sense (External image)
  * Meditation of the senses (A sound)
  * Open monitoring (Mindfulness)
  Arms: Nurses receiving mindfulness meditation

SUMMARY:
Background: Nurses have experienced several stressors, the most important of which are increased workloads, long shifts, patients' negative results, some patients not responding to treatment, death at high rates, late detection of disease cases, lack of social support system, and limited typical coping.

Aim: The purpose of this study is to assess the effectiveness of mindfulness meditation for clinical nurses to improve perceived stress and somatic symptoms and pro-inflammatory factors. Among Jordanian clinical nurses.

Methodology: The study will be conducted using a post-test randomized controlled experimental design. The study data will be collected using a self-report questionnaire and blood sampling from 102 nurses in in King Abdullah hospitals at baseline and at the end of intervention. Data were analyzed using the Statistical Package for Social Science (SPSS), Version 26.

DETAILED DESCRIPTION:
Introduction

The nursing profession has historically been associated with significant chronic stress due to frequent exposure to various work-related stressors. These include psychological or physical violence in the workplace, coping with patient deaths, staff shortages, and a high patient load. The pandemic has added additional pressures and stressors, including dealing with emergency patients, fear of exposure to the virus, increased working hours, imbalance between work and personal life, disruption of family life, and inability to adapt to a rapidly changing work environment. These unprecedented situations require nurses to work long hours with more limited resources, which lead to sever level of chronic stress.

Some nurses demonstrate resilience in the face of stress. However, most experience prolonged stress that dysregulate physiological functions and reduce physical and psychological health. According to Yaribeygi, et al. (2017) psychological stress is associated with the activation of several body systems, including the hypothalamic pituitary-adrenal axis and the sympathetic nervous system. The activation of these two pathways results in elevated cortisol and catecholamines. Although the mechanism is still not fully understood, chronic stress results in prolonged, excessive production of cortisol, causing chronic release of pro-inflammatory factors such as InterLeukine-6 (IL-6) and TNFα. Such a chronic increase of proinflammatory markers in healthy individuals is generally known as low-grade inflammation, which is associated to several chronic illness such as cardiovascular disease, type 2 diabetes, metabolic syndrome and major depression. Studies have revealed that persistent workplace stress lead to increased inflammatory activity in healthcare professionals with unsatisfied working conditions.

The elevated cortisol and catecholamines also puts nurses at increased risk of developing somatic symptoms, known as physical complaints, that cannot be explained by medical condition, mental disorder, or substance abuse. These complaints are often associated with psychological stress and may involve sleep problems, digestive problems, heart disease, palpitations, headache, weight gain and memory and concentration and muscle tension. A recent systematic review investigating the prevalence of somatic symptoms during the COVID-19 pandemic showed that such symptoms, including shortness of breath, dyspnea, palpitations, and pain, were reported by 7.4% to 67% of patients, healthcare workers, and the general population. Also, a study revealed that the overall prevalence rates somatic symptoms among nurses during COVID-19 pandemic was 50%. Such symptoms affect negatively nurses' quality of life and job performance, resulting in increased errors in patient care.

The high prevalence of somatic symptoms and low-grade inflammation among healthcare professionals, including nurses, indicates unmet needs within this population. Addressing these needs requires implementing preventive strategies to enhance mental resilience, particularly for high-risk individuals such as nurses. Mindfulness is one of the most important methods used in psychotherapy, which is strongly associated with promotion physical and psychological well-being, it is an effective method for reducing stress and improving health. The practice of mindfulness originally began in Asian culture due to meditative practices in Buddhist philosophy and eastern spiritual traditions; where it emphasized the value of presence, non-exaggeration, and experience acceptance. In the 1970s and 1980s, mindfulness began to be used in Western countries, and it gradually developed into one of the most important techniques in contemporary psychotherapy. In recent years, the practice of mindfulness has been widely applied in both clinical and non-clinical settings

. Several studies support the potential benefits of MBI on psychological health among nurses. Duarte and Pinto-Gouveia reported that an abbreviated MBI resulted in significant improvement in compassion fatigue, burnout, stress, life satisfaction and self-compassion in oncology nurses. In a systematic review conducted by Chiappetta et al., MBI has been found to significantly decrease stress, burnout, anxiety, and depression, and improve self-compassion and quality of life among healthcare professionals. Similarly, Lomas et al. in their systematic review supported these results, indicating that MBI significantly reduced anxiety, depression, stress, and overall well-being in nurses. Lin et al. conducted in randomized control trial and found that an eight-week MBSR program reduced stress and negative affect while increasing positive affect and resilience among Chinese nurses. Two other systematic review studies by Sulosaari et al. and Ramachandran et al. found that MBI significantly improved psychological well-being, resilience, and quality of life, while reducing stress, depression, and burnout among nurses.

However, rare studies examined the effect of such intervention on nurses' physical health such as somatic symptoms and inflammation. MBI, as a holistic approach, has been found to improve a wide range of health outcomes in different healthy and ill populations including somatic symptoms and proinflammatory markers. The mechanism underlying the effect of mindfulness intervention on somatic symptoms and inflammatory biomarkers can be explained by the Cognitive Reappraisal Model. According to this model, the effects of mindfulness practices on health outcomes are postulated to be mediated by improvement in trait mindfulness and emotion regulation skills. Frequent mindfulness practice boosts the mental capacity of mindfulness trait, known as present-moment awareness and non-judgmental observation over thought and feelings. Such mental capacity helps people become aware of and detach from the stressful thoughts and emotions by enabling cognitive reappraisal as an emotion regulation skill. This is the process by which people can re-interpret stressful events in less negative ways, resulting in lower perceived stress levels. By alleviating perceived stress through cognitive reappraisal, mindfulness intervention can improve the physiological responses associated with stress, such as the activation of the hypothalamic-pituitary-adrenal (HPA) axis and the release of proinflammatory biomarkers.

Research have supported the hypotheses of the Cognitive Reappraisal Model indicating the mindfulness intervention can potentially reduce somatic symptoms and inflammatory biomarkers (e.g. interleukin 6 and TNF-alpha) by reducing perceived stress. However, to the best of our knowledge, these effects have not been examined among nurses in Jordan. Thus, this study aimed to examine the effect of mindfulness intervention on perceived stress, somatic symptoms, proinflammatory biomarkers such as interleukin 6 and TNF alpha.

Methods Design This was an experimental study using pretest post-test randomized controlled design. This design is described as a plausible tool in terms of the control on extraneous variables using various strategies, including manipulation, control group, and random assignment. Participants were randomly assigned into the experimental and control groups. Researchers who are not involved in the recruitment process and patient assessment, were randomly assign the participants to the intervention group or the control group, using a simple 1:1 computer-generated sequence.

Sample and setting The hospital can accommodate 750 beds, but in an emergency, that number may be raised to 900. Participants who were having psychiatric illnesses, disorders of the immune system (e.g., immunodeficiency or autoimmune disorders), and current infections and taking anti-inflammatory or antimicrobial medications were excluded.

G*Power software version 3.1 was used to calculate the required sample size. Based on an independent t-test, with an alpha level of 0.05, a power of 0.8, and a moderate effect size of 0.5, the required sample size was determined to be 102 participants.

Intervention The experimental group received eight 60-minute weekly sessions of MBI over eight weeks in a private and quiet room at the hospital, according to Smith's (2005) recommendation. The study intervention was an audio based MBI sent to them by the WhatsApp application. It is a free, self-paced program developed by a study researcher based on the Smith's (2005) protocol. This study researcher was an experienced practitioner with a Ph.D. degree in nursing and received extensive stress management training, including MBI at a Psychology Department at a university in the United States 10 years ago. Since then, he has been practicing the MBI daily. The audio recording of the MBI was evaluated and validated for the clarity of voice and the MBI content by two psychologists who are experts in MBI.

However, these eight weekly sessions were conducted by one of the study researchers to explain the rationale and procedures of MBI including a demonstration of the entire MBI protocol for the participants in the experimental group. He was also present during the delivery of MBI session to confirm and facilitate the administration of the MBI sessions and answer any participants' questions. This study researcher has a master's degree in nursing and received extensive MBI training. The participants in the experimental groups were encouraged not to share any information regarding the MBI with anyone during the study.

The theory-based program (Smith, 2005) includes the ABC standardized versions of MBI (Smith, 2005), described as follows:

* Meditation of the body (Body sense meditation): Individuals pay attention in the present moment without judgment.
* Meditation of the body (Rocking meditation): Individuals allow themselves to gently rock back and forth in their chairs, effortlessly and quietly, while paying mindful attention to the gentle, silent motion of the rocking
* Meditation of the body (Breathing meditation): Individuals allow their breathing to flow naturally, free and easy, while simply focusing on the rhythm of the breath as it moves in and out.
* Meditation of mind (Mentra meditation): Individuals allow a calming word, like 'peace,' to gently enter their minds, like an echo in the distance, while quietly and effortlessly focusing as the word repeats over and over
* Meditation of mind (visual Image): Individuals visualize a simple spot of light, such as a candle flame or a star, and quietly focus their attention on it.
* Meditation of sense (External image): Individuals slowly open their eyes halfway and gently gaze at a certain object (e.g. candle) in front of them
* Meditation of the senses (A sound): Individuals choose a quiet, continuous sound and gently focus their attention on it
* Open monitoring (Mindfulness): Nurses quietly observe, acknowledge, and release every internal and external stimulus-such as thoughts, feelings, sensations, sounds, and ideas-that enters their awareness. They refrain from analyzing, resisting, or trying to manage these experiences and do not concern themselves with the connections between each stimulus. Instead, they simply allow each stimulus to arise and fade away, patiently waiting for the next one.

Participants in the control group were not asked to do anything during the study, except their traditional practices. However, mindfulness meditation was provided to them after the study.

Data collection and Ethical consideration Following IRB approval, one of the study researchers contacted the hospital administrators to seek permission to conduct the study. Once approval was granted, the nurses were approached in person, and the study's purpose was explained to them. Those who agreed to participate were asked to sign a consent form. Participants' confidentiality and anonymity were strictly maintained. A researcher not involved in recruitment or patient assessment then randomly assigned participants to either the intervention or control group using a simple 1:1 computer-generated sequence. The mindfulness-based intervention (MBI) schedule was provided to participants in the experimental group, aligned with their work schedules.

Baseline and post-intervention measurements were conducted at the hospital by a researcher (nurse). To minimize measurement errors due to variations in data collection, self-reported measures were completed after the objective measures, such as biological markers, to reduce stress-related biases. All measurements for both the intervention and control groups were taken under consistent conditions, including room temperature and environment, by a well-trained nurse with a master's degree in nursing. The ELISA protocol for blood sampling was meticulously followed, and neurotransmitter and hormone levels were measured at 8 a.m. for all participants, who were seated during testing.

Statistical Analysis Data were analyzed using the Statistical Package for Social Science (SPSS), Version 26. Descriptive statistics were used to describe the study participants as appropriate. For instance, frequency and percentage were used to describe the categorical variables, while mean and standard deviation (SD) were used to describe the continuous variables. Also, the baseline statistical equivalence between the study groups on the dependent and sociodemographic variables was evaluated using independent t-tests. Dependent t-tests were used to examine if there were statistically significant changes between the pretest and posttest in each study group. Finally, independent t-tests were used to examine if there was a statistically significant difference between the experimental and control group at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Nurse working in the hospital in Jordan
* Being at least 21 years old
* Having a smartphone
* Being able to read and write in English

Exclusion Criteria:

* Having psychiatric illnesses
* Having disorders of the immune system (e.g., immunodeficiency or autoimmune disorders) and current infections.
* Taking anti-inflammatory or antimicrobial medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Mindful Attention Awareness Scale | From enrollment to the end of intervention at 8 weeks
  Mindful Attention Awareness Scale (MAAS) (Brown & Ryan, 2003) was used to measure dispositional mindfulness.
  It is one-dimensional scale including 15 items measured on a six-point likert type scale, ranging from 1 (almost always) to 6 (almost never). The score range is between 15 and 90, with higher score indicting higher levels of mindfulness. The scale has shown strong psychometric properties when validated in college students. It showed single-factor construct in MAAS structure and a Chronbach's alpha of 0.82 in university sample. Correlational, quasi-experimental, and laboratory studies have shown that the MAAS taps a unique quality of consciousness that is related to, predictive of, a variety of self-regulation and well-being constructs. The Arabic version showed acceptable levels of validity and reliablity in an Arab population and nursing students.
Perceived Stress Scale | From enrollment to the end of intervention at 8 weeks
  The Perceived Stress Scale (PSS) is used to measure the degree to which situations in one's life are appraised as stressful (unpredictable, uncontrollable, and overloaded). It composes of 10 items rated on a 5-point Likert scale (0=never, 4= very often), which are relatively free of content specific to any subpopulation group. The total scores of the scale range from 0 to 40, with higher scores indicating higher levels of perceived stress (Cohen et al., 1983). PSS has been validated among college students. Internal consistency coefficients for the PSS ranged from .84 to 36, and test- retest reliability was .85 (Cohen et al., 1983). The Arabic version of the scale demonstrated an acceptable level of reliability and validity among Arabic adult population (Almadi, et al., 2012).
The Patient Health Questionnaire-15 | From enrollment to the end of intervention at 8 weeks
  The The Patient Health Questionnaire-15 (PHQ-15) is a self-reported somatic symptoms subscale, derived from the full Patient-Health-Questionnaire (Spitzer, et al., 1999; Löwe, Zipfel, Herzog, 2002; Kroenke et al., 2002). It is a 15-item instrument that assesses 15 common somatic symptoms. Subjects were asked to rate the severity of symptoms as 0 ("not bothered at all"), 1 ("bothered a little"), or 2 ("bothered a lot"). The score ranges from 0 to 30 and scores of ≥5, ≥10, ≥15 represent mild, moderate and severe levels of somatization respectively. Evidence supports reliability and validity of the PHQ-15 as a measure of physical symptoms in the general population. The scores of the PHQ-15 were highly correlated with the scores of depressions and the physical component summary scale of health-related quality of life (Kocalevent, Hinz, &Brähler, 2013). The internal consistency (Cronbach's α) for the PHQ-15 was 0.82 (Kocalevent, Hinz, & Brähler, 2013).
Change in serum levels of inflammatory biomarkers (Leptin, IL-6, TNF-α) as measured by ELISA | From enrollment to the end of intervention at 8 weeks
  The blood sampling and analysis protocol for inflammatory biomarkers (leptin, IL-6, and TNF-α) was rigorously followed using the ELISA technique. Blood samples were collected via venipuncture, stored at 4°C, and processed within two hours to maintain integrity. Plasma or serum was separated by centrifugation and stored at -80°C until analysis. Biomarker levels were quantified in ng/mL for leptin and pg/mL for IL-6 and TNF-α, following specific ELISA procedures. Elevated levels of these biomarkers indicate increased low-grade inflammation. Overall, the analysis reflects systemic inflammation and aids in assessing patients' inflammatory status.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Alhawatmeh, Doctoral degree, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- King Abdullah University Hospital, Irbid, None Selected, Jordan

IPD SHARING:
Plan to Share IPD: No
Due to the ethical constraints

REFERENCES:
- [Result] Rayan A, Ahmad M. The psychometric properties of the mindful attention awareness scale among Arab parents of children with autism spectrum disorder. Arch Psychiatr Nurs. 2018 Jun;32(3):444-448. doi: 10.1016/j.apnu.2018.01.001. Epub 2018 Jan 3. PMID 29784228
- [Result] Alhawatmeh HN, Rababa M, Alfaqih M, Albataineh R, Hweidi I, Abu Awwad A. The Benefits of Mindfulness Meditation on Trait Mindfulness, Perceived Stress, Cortisol, and C-Reactive Protein in Nursing Students: A Randomized Controlled Trial. Adv Med Educ Pract. 2022 Jan 13;13:47-58. doi: 10.2147/AMEP.S348062. eCollection 2022. PMID 35046747
- [Result] Geiger PJ, Boggero IA, Brake CA, Caldera CA, Combs HL, Peters JR, Baer RA. Mindfulness-Based Interventions for Older Adults: A Review of the Effects on Physical and Emotional Well-being. Mindfulness (N Y). 2016 Apr;7(2):296-307. doi: 10.1007/s12671-015-0444-1. Epub 2015 Sep 14. PMID 27200109
- [Result] Carlson LE. Mindfulness-based interventions for physical conditions: a narrative review evaluating levels of evidence. ISRN Psychiatry. 2012 Nov 14;2012:651583. doi: 10.5402/2012/651583. Print 2012. PMID 23762768
- [Result] Theocharis A, Antonopoulos V, Christodoulou NG. Somatic symptoms associated with mental distress during the COVID-19 pandemic: a systematic review. Australas Psychiatry. 2023 Apr;31(2):147-156. doi: 10.1177/10398562231156380. Epub 2023 Feb 24. PMID 36825513
- [Result] Kaltenegger HC, Weigl M, Becker L, Rohleder N, Nowak D, Quartucci C. Psychosocial working conditions and chronic low-grade inflammation in geriatric care professionals: A cross-sectional study. PLoS One. 2022 Sep 15;17(9):e0274202. doi: 10.1371/journal.pone.0274202. eCollection 2022. PMID 36107874
- [Result] Furman D, Campisi J, Verdin E, Carrera-Bastos P, Targ S, Franceschi C, Ferrucci L, Gilroy DW, Fasano A, Miller GW, Miller AH, Mantovani A, Weyand CM, Barzilai N, Goronzy JJ, Rando TA, Effros RB, Lucia A, Kleinstreuer N, Slavich GM. Chronic inflammation in the etiology of disease across the life span. Nat Med. 2019 Dec;25(12):1822-1832. doi: 10.1038/s41591-019-0675-0. Epub 2019 Dec 5. PMID 31806905
- [Result] Roenneberg, T., et al. (2019). A practical tool to assess circadian disruption: The Social Jetlag Questionnaire. Chronobiology International, 36(6), 830-838.
- [Result] Mehling W. Differentiating attention styles and regulatory aspects of self-reported interoceptive sensibility. Philos Trans R Soc Lond B Biol Sci. 2016 Nov 19;371(1708):20160013. doi: 10.1098/rstb.2016.0013. Epub 2016 Oct 10. PMID 28080970
- [Result] Pan X, Xiao Y, Ren D, Xu ZM, Zhang Q, Yang LY, Liu F, Hao YS, Zhao F, Bai YH. Prevalence of mental health problems and associated risk factors among military healthcare workers in specialized COVID-19 hospitals in Wuhan, China: A cross-sectional survey. Asia Pac Psychiatry. 2022 Mar;14(1):e12427. doi: 10.1111/appy.12427. Epub 2020 Oct 21. PMID 33089622
- [Result] Micheli N, Porcelli P, Barrault-Couchouron M, Dantzer C. Does the practice of mindfulness reduce somatic symptoms and COVID-19-related anxiety? A community-based survey. Front Psychol. 2022 Dec 9;13:996559. doi: 10.3389/fpsyg.2022.996559. eCollection 2022. PMID 36571039
- [Result] Starc J. Stress Factors among Nurses at the Primary and Secondary Level of Public Sector Health Care: The Case of Slovenia. Open Access Maced J Med Sci. 2018 Feb 10;6(2):416-422. doi: 10.3889/oamjms.2018.100. eCollection 2018 Feb 15. PMID 29531616
- [Result] Sulosaari V, Unal E, Cinar FI. The effectiveness of mindfulness-based interventions on the psychological well-being of nurses: A systematic review. Appl Nurs Res. 2022 Apr;64:151565. doi: 10.1016/j.apnr.2022.151565. Epub 2022 Jan 15. PMID 35307128
- [Result] Lin L, He G, Yan J, Gu C, Xie J. The Effects of a Modified Mindfulness-Based Stress Reduction Program for Nurses: A Randomized Controlled Trial. Workplace Health Saf. 2019 Mar;67(3):111-122. doi: 10.1177/2165079918801633. Epub 2018 Oct 29. PMID 30370837
- [Result] Lomas T, Medina JC, Ivtzan I, Rupprecht S, Eiroa-Orosa FJ. A systematic review of the impact of mindfulness on the well-being of healthcare professionals. J Clin Psychol. 2018 Mar;74(3):319-355. doi: 10.1002/jclp.22515. Epub 2017 Jul 28. PMID 28752554
- [Result] Nourian M, Nikfarid L, Khavari AM, Barati M, Allahgholipour AR. The Impact of an Online Mindfulness-Based Stress Reduction Program on Sleep Quality of Nurses Working in COVID-19 Care Units: A Clinical Trial. Holist Nurs Pract. 2021 Sep-Oct 01;35(5):257-263. doi: 10.1097/HNP.0000000000000466. PMID 34407023
- [Result] Dundas I, Thorsheim T, Hjeltnes A, Binder PE. Mindfulness Based Stress Reduction for Academic Evaluation Anxiety: A Naturalistic Longitudinal Study. J College Stud Psychother. 2016 Apr 2;30(2):114-131. doi: 10.1080/87568225.2016.1140988. Epub 2016 Apr 13. PMID 27227169
- [Result] Bartlett L, Buscot MJ, Bindoff A, Chambers R, Hassed C. Mindfulness Is Associated With Lower Stress and Higher Work Engagement in a Large Sample of MOOC Participants. Front Psychol. 2021 Sep 10;12:724126. doi: 10.3389/fpsyg.2021.724126. eCollection 2021. PMID 34566805
- [Result] Sheng JA, Bales NJ, Myers SA, Bautista AI, Roueinfar M, Hale TM, Handa RJ. The Hypothalamic-Pituitary-Adrenal Axis: Development, Programming Actions of Hormones, and Maternal-Fetal Interactions. Front Behav Neurosci. 2021 Jan 13;14:601939. doi: 10.3389/fnbeh.2020.601939. eCollection 2020. PMID 33519393
- [Result] Yaribeygi H, Panahi Y, Sahraei H, Johnston TP, Sahebkar A. The impact of stress on body function: A review. EXCLI J. 2017 Jul 21;16:1057-1072. doi: 10.17179/excli2017-480. eCollection 2017. PMID 28900385
- [Derived] Alhawatmeh H, Abusaif L, Alharrasi M, Abuhammad S. Impact of Mindfulness Meditation on Perceived Stress, Somatic Symptoms and Inflammatory Biomarkers Among Clinical Nurses. J Nurs Scholarsh. 2026 Jan;58(1):e70067. doi: 10.1111/jnu.70067. PMID 41580885